CLINICAL TRIAL: NCT01484977
Title: Open-label, Single Arm, Study Evaluating Tolerability and Efficacy of Lacosamide When Added to Levetiracetam With Withdrawal of Concomitant Sodium Channel Blocking Antiepileptic Drug in Subjects With Uncontrolled Partial-onset Seizures
Brief Title: eValuation of the Efficacy and toleRability of Vimpat When Added to lEvetiracetam
Acronym: VERVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0980; 2011-002461-37 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: Lacosamide; Epilepsy; Levetiracetam; Sodium Channel Blockers
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Lacosamide will be added to levetiracetam while withdrawing the sodium channel blocking antiepileptic drug (AED)
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — 50 mg and 100 mg lacosamide tablets will be combined and taken in two equal doses per day to provide the required total daily dosage of 100 - 600 mg/day. Subjects were titrated to a minimum of 200 mg/ day during the Treatment Period.
  Maximum duration of study drug administration is approximately 23 weeks.
  Other Names: VIMPAT®; SPM927; Harkoseride

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of the study drug lacosamide (200-600 mg/day) when added to a stable dose of levetiracetam (1000-3000 mg/day) with withdrawal of the concomitant sodium channel blocking-antiepileptic drug (AEDs) in subjects not well controlled on their current regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, at least 18 years of age
* Subject has a diagnosis of epilepsy with partial-onset seizures according to the International Classification of Epileptic Seizures (1981)
* Subject is taking levetiracetam (LEV) in combination with 1 sodium channel blocking antiepileptic drug (defined as carbamazepine, lamotrigine, oxcarbazepine, phenytoin, or eslicarbazepine) as adjunctive treatment for epilepsy
* The minimum required seizure frequency during the 8-week Retrospective Seizure Baseline is on average ≥ 2 partial-onset seizures per 28 days with at least 1 seizure per 4 week period within the 8-week Retrospective Seizure Baseline. Additionally, subjects must experience at least 1 seizure during the 4-week Prospective Seizure Baseline
* Subject has been maintained on a stable dose of LEV and a sodium channel blocking antiepileptic drug (SCB-AED) for at least 4 weeks prior to the Screening Visit (Visit 1) and during the 4-week Prospective Seizure Baseline
* The minimum required seizure frequency during the 8-week Retrospective Seizure Baseline is on average ≥ 2 partial-onset seizures per 28 days (based on investigator assessment of subject report) with at least 1 seizure per 4 week period within the 8-week Retrospective Seizure Baseline
* Subject has been maintained on a stable dose of levetiracetam (LEV) and a sodium channel blocking antiepileptic drug (SCB-AED) for at least 4 weeks prior to the Screening Visit (Visit 1) and during the 4-week Prospective Seizure Baseline, with or without additional concurrent stable vagal nerve stimulation (VNS). The VNS must have been in place for at least 6 months prior to the Screening Visit (Visit 1) with constant settings for at least 4-weeks prior to the Screening Visit (Visit 1) and throughout the duration of the study

Exclusion Criteria:

* Previous use of lacosamide
* History of alcohol or drug abuse
* History of seizure disorder characterized primarily by isolated auras
* History of primary generalized seizures
* History of status epilepticus within the 12-months
* History of clustering seizures
* Nonepileptic events, including pseudoseizures that could be confused with seizures
* History of any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in this study
* Lifetime history of suicide attempt, or suicidal ideation in the past 6 months
* Hypersensitivity to any component of lacosamide (LCM)
* History of acute or sub-acute progressive central nervous system disease
* History of severe anaphylactic reaction or serious blood dyscrasias
* Impaired renal function (ie, Creatinine Clearance (CLcr) is lower than 30 mL/min) at Visit 1
* History of sick sinus syndrome without a pacemaker, or atrioventricular (AV) block, or subject has any other clinically significant electrocardiogram (ECG) abnormalities
* History sodium channelopathy, such as Brugada syndrome
* History of myocardial infarction in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 877-822-9493
Locations (54):
- United States (30):
  - 110, Huntsville, Alabama
  - 004, Phoenix, Arizona
  - 001, Fresno, California
  - 008, Orange, California
  - 030, Oxnard, California
  - 108, Sacramento, California
  - 025, Bradenton, Florida
  - 015, Ocala, Florida
  - 049, Panama City, Florida
  - 114, Port Charlotte, Florida
  - 012, Sarasota, Florida
  - 014, Tampa, Florida
  - 003, Wellington, Florida
  - 123, Louisville, Kentucky
  - 006, Hammond, Louisiana
  - 112, Waldorf, Maryland
  - 129, Golden Valley, Minnesota
  - 023, Springfield, Missouri
  - 088, Missoula, Montana
  - 020, Camden, New Jersey
  - 131, Greensboro, North Carolina
  - 002, Akron, Ohio
  - 027, Canton, Ohio
  - 022, Columbus, Ohio
  - 005, Dayton, Ohio
  - 013, Oklahoma City, Oklahoma
  - 028, Lubbock, Texas
  - 017, Salt Lake City, Utah
  - 139, Madison, Wisconsin
  - 024, Milwaukee, Wisconsin
- Australia (2):
  - 075, Chatswood
  - 079, Parkville
- Bulgaria (5):
  - 036, Rousse
  - 037, Sofia
  - 080, Sofia
  - 081, Sofia
  - 082, Sofia
- Denmark (2):
  - 059, Aarhus
  - 087, Copenhagen
- France (3):
  - 042, Angers
  - 040, Limoges
  - 046, Paris
- Germany (3):
  - 065, Bielefeld
  - 066, Hamburg
  - 068, Tübingen
- Romania (5):
  - 096, Bucharest
  - 099, Bucharest
  - 097, Lasi
  - 038, Târgu Mureş
  - 095, Târgu Mureş
- Spain (3):
  - 051, Manresa
  - 053, Oviedo
  - 050, Seville
- 102, Gothenburg, Sweden

REFERENCES:
- [Result] Baulac M, Byrnes W, Williams P, Borghs S, Webster E, De Backer M, Dedeken P. Lacosamide and sodium channel-blocking antiepileptic drug cross-titration against levetiracetam background therapy. Acta Neurol Scand. 2017 Apr;135(4):434-441. doi: 10.1111/ane.12691. Epub 2016 Oct 6. PMID 27714769
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment for the SP0980 study began in December 2011. It concluded in January 2014. This was a multicenter study with subjects enrolled by 30 sites across North America, 12 in Western Europe, 10 in Eastern Europe, and 2 in Oceania.
Pre-assignment Details: The participant flow consists of subjects in the Safety Set (SS). The SS is all subjects who received at least 1 dose of lacosamide.
Groups:
- Lacosamide: Lacosamide will be added to levetiracetam while withdrawing the sodium channel blocking antiepileptic drug (AED).
  Lacosamide: 50 mg and 100 mg lacosamide tablets will be combined and taken in two equal doses per day to provide the required total daily dosage of 100 - 600 mg/day. Subjects were titrated to a minimum of 200 mg/ day during the Treatment Period.
  Maximum duration of study drug administration is approximately 23 weeks.
Period: Overall Study
Arm/Group | Lacosamide
Started | 120
Completed | 93
Not Completed | 27
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 4
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Subject Protocol Non-compliant | 1
Not completed — Moving Overseas | 1
Not completed — Low White Blood Cell Count | 1
Not completed — Lack of Compliance | 1

BASELINE CHARACTERISTICS:
Population: The Baseline characteristics consist of subjects in the Safety Set (SS). The SS is all subjects who received at least 1 dose of lacosamide.
Arm/Group | Lacosamide
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 114
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 46
Weight [Mean (Standard Deviation); unit: kilograms] | 76.39 (19.98)
Height [Mean (Standard Deviation); unit: centimeters] | 168.02 (10.55)
BMI [Mean (Standard Deviation); unit: kilogram/ square meter] | 27.00 (6.45)
Racial Group [Number; unit: participants]
  American Indian/Alaskan Native | 1
  Asian | 3
  Black | 8
  Native Hawaiian or other Pacific Islander | 0
  White | 96
  Other/Mixed | 12
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 103

OUTCOME MEASURES:

1. Primary Outcome: Retention at the End of the 21-week Treatment Period
Description: Retention is a summary measure that integrates both the patient's and clinician's assessment of efficacy and tolerability in epilepsy clinical studies to provide a measure of effectiveness.
Time Frame: Duration of the Treatment Period (21 Weeks)
Population: The primary analysis consists of subjects in the Safety Set (SS). The SS is all subjects who received at least 1 dose of lacosamide.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 120
percentage of participants | 73.3
Statistical Analysis 1: Comparison: Lacosamide; Analyses of the primary efficacy variable will be descriptive only. No hypothesis tests are planned. The number and percentage of subjects remaining in the study through the 21-Week Treatment Period will be calculated. Subjects with retention will be counted in the numerator. All subjects in the relevant population will be used as the denominator. This percentage will be known as the retention rate, along with the 95 % confidence interval based on the normal approximation; Test type: Superiority or Other; Retention Rate = 73.3, 95% CI 2-sided [65.42 to 81.25]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were recorded during the course of the SP0980 study, which began in December 2011 and concluded in January 2014.
Description: TEAE reporting refers to the Safety Set (SS). The SS is all subjects who received at least 1 dose of lacosamide.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 8/120
Other Adverse Events (participants affected / at risk) | 52/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=120)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vulvovaginitis Trichomonal (Infections and infestations) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Asthma (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=120)
Nausea (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 10 (13)
Dizziness (Nervous system disorders) | 28 (40)
Headache (Nervous system disorders) | 18 (21)
Convulsion (Nervous system disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.